CLINICAL TRIAL: NCT06898931
Title: A Study of Language Intervention Training for Cognitive Protection in High-risk Cardio-Cerebrovascular Elderly Population
Brief Title: Language Intervention Training for Cognitive Protection in High-risk Cardio-Cerebrovascular Elderly Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Min Lou, Prof, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Boost
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Vascular Cognitive Impairment No Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rountine (No Intervention): The control group will not receive any language intervention training and will maintain their usual daily routines.
- Dialect Interpreting Training (Experimental): The intervention group will receive a combination of offline and online language-switching training. The offline intervention will last for 2 months, with three training sessions per week, each lasting 1 hour. The training content will simulate the interpreting process, requiring participants to switch and convert rapidly and accurately between two dialects, covering multiple aspects including listening comprehension, oral expression, and information processing. The online intervention will last for 4 months, during which participants will regularly complete exercises through a language training app or website and upload their assignments.
  Interventions: Behavioral: Dialect Interpreting Training

INTERVENTIONS:
Behavioral: Dialect Interpreting Training — The intervention group will receive a combination of offline and online language-switching training. The offline intervention will last for 2 months, with three training sessions per week, each lasting 1 hour. The training content will simulate the interpreting process, requiring participants to switch and convert rapidly and accurately between two dialects, covering multiple aspects including listening comprehension, oral expression, and information processing. The online intervention will last for 4 months, during which participants will regularly complete exercises through a language training app or website and upload their assignments.
  Arms: Dialect Interpreting Training

SUMMARY:
The global population is aging rapidly, with the number of elderly people with dementia projected to rise sharply, posing significant challenges to quality of life and societal burden.Frequent language switching, such as in interpreting, enhances cognitive abilities by improving attention, flexibility, and memory.Dialect-switching training, similar to interpreting, is a non-invasive method that shows potential for promoting cognitive health in the elderly but remains under-researched.This study aims to investigate the cognitive-enhancing effects of a dialect-switching training program on older adults with vascular risk factors through a six-month intervention.

DETAILED DESCRIPTION:
The global population is aging rapidly, with those aged 65+ expected to reach 16% of the total population by 2050. Aging is linked to increased cognitive impairment risks, including dementia prevalence rates of 5%-10% among the elderly in developed countries. In China, the number of elderly with dementia is projected to soar from 7.4 million to 18 million by 2030 without intervention. This trend poses significant challenges to quality of life and societal burden.

Language experiences, particularly frequent switching between languages, enhance cognitive abilities. Interpreting, which demands high-intensity language switching, significantly improves cognitive control and memory. Interpreters' need for rapid language conversion and reliance on attention, flexibility, and inhibition contribute to their cognitive advantages.

Similar to interpreting, switching between dialects and standard language requires high-frequency, high-intensity language conversion. This non-invasive training method is suitable for promoting cognitive health in the elderly. However, its potential benefits for cognitive enhancement in this population remain underexplored.

This study aims to design a dialect-switching training program simulating interpreting and investigate its potential cognitive-enhancing effects through a six-month intervention in older adults with vascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 60 years
* High risk of stroke (with ≥ 3 of 8 stroke risk factors, including hypertension, dyslipidemia, diabetes, atrial fibrillation or valvular heart disease, smoking history, obvious overweight or obesity, lack of exercise, family history of stroke, or with transient ischemic attack)
* command of Hangzhou dialect
* Written informed consent available
* Willingness to complete all assessments and participate in follow-up
* Adequate Visual and auditory acuity to undergo neuropsychological testing

Exclusion Criteria:

* previously diagnosed dementia
* Suspected dementia after clinical assessment by study physician at screening visit
* Previous history of major head trauma and any intracranial surgery
* Intracranial abnormalities, such as intracerebral hemorrhage, subarachnoid hemorrhage and other space occupying lesions
* Extrapyramidal symptoms or mental illness which may affect neuropsychological measurement
* Severe loss of vision, hearing, or communicative ability
* Patients presenting a malignant disease with life expectancy < 3 years
* Participation in an ongoing investigational drug study
* Any MRI contraindications

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Changes in brain functional network connectivity assessed by resting state functional magnetic resonance imaging (fMRI) | 6 months
  Primary Outcome

SECONDARY OUTCOMES:
Changes in brain functional network efficiency assessed by resting state fMRI | 2 years
  long-term secondary outcome
Changes in brain functional network activity intensity assessed by resting state fMRI | 2 years
  long-term secondary outcome
Changes in brain functional network efficiency assessed by resting state fMRI | 5 years
  long-term secondary outcome
Changes in brain functional network activity intensity assessed by resting state fMRI | 5 years
  long-term secondary outcome
Changes in brain functional network efficiency assessed by resting state fMRI | 6 months
  short-term secondary outcome
Changes in brain functional network activity intensity assessed by resting state fMRI | 6 months
  short-term secondary outcome
Changes in brain functional network connectivity assessed by resting state fMRI | 2 years
  long-term secondary outcome
Changes in brain functional network connectivity assessed by resting state fMRI | 5 years
  long-term secondary outcome
Global cognitive function change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network (NINDS-CSN) protocol (higher scores mean a better outcome) | 6 months
  short-term secondary outcome
Global cognitive function change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network (NINDS-CSN) protocol (higher scores mean a better outcome) | 2 years
  long-term secondary outcome
Global cognitive function change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network (NINDS-CSN) protocol (higher scores mean a better outcome) | 5 years
  long-term secondary outcome
Cognitive domain change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network (NINDS-CSN) protocol (higher scores mean a better outcome) | 6 months
  short-term secondary outcome
Cognitive domain change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network (NINDS-CSN) protocol (higher scores mean a better outcome) | 2 years
  long-term secondary outcome
Cognitive domain change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network (NINDS-CSN) protocol (higher scores mean a better outcome) | 5 years
  long-term secondary outcome
Cognitive function change assessed with Mini-Mental State Examination (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 6 months
  short-term secondary outcome
Cognitive function change assessed with Mini-Mental State Examination (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 2 years
  long-term secondary outcome
Cognitive function change assessed with Mini-Mental State Examination (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 5 years
  long-term secondary outcome
Cognitive function change assessed by Montreal Cognitive Assessment (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 6 months
  short-term secondary outcome
Cognitive function change assessed by Montreal Cognitive Assessment (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 2 years
  long-term secondary outcome
Cognitive function change assessed by Montreal Cognitive Assessment (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 5 years
  long-term secondary outcome
Changes in white matter hyperintensity (WMH) assessed on MRI with T2-Fluid-Attenuated-Inversion-Recovery (FLAIR) sequence | 6 months
  short-term secondary outcome
Changes in lacunes assessed on MRI with T2 FLAIR sequence | 6 months
  short-term secondary outcome
Changes in perivascular spaces assessed on MRI with T2 FLAIR sequence | 6 months
  short-term secondary outcome
Changes in microbleeds assessed on MRI with Susceptibility Weighted Imaging (SWI) sequence sequence | 6 months
  short-term secondary outcome
Changes in brain atrophy (width of the sulci greater than 5mm) assessed on MRI | 6 months
  short-term secondary outcome
Changes in white matter hyperintensity (WMH) assessed on MRI with T2 FLAIR sequence | 2 years
  long-term secondary outcome
Changes in white matter hyperintensity (WMH) assessed on MRI with T2 FLAIR sequence | 5 years
  long-term secondary outcome
Changes in lacunes assessed on MRI with T2 FLAIR sequence | 2 years
  long-term secondary outcome
Changes in lacunes assessed on MRI with T2 FLAIR sequence | 5 years
  long-term secondary outcome
Changes in perivascular spaces assessed on MRI with T2 FLAIR sequence | 2 years
  long-term secondary outcome
Changes in perivascular spaces assessed on MRI with T2 FLAIR sequence | 5 years
  long-term secondary outcome
Changes in microbleeds assessed on MRI with SWI sequence sequence | 2 years
  long-term secondary outcome
Changes in microbleeds assessed on MRI with SWI sequence sequence | 5 years
  long-term secondary outcome
Changes in brain atrophy (width of the sulci greater than 5mm) assessed on MRI | 2 years
  long-term secondary outcome
Changes in brain atrophy (width of the sulci greater than 5mm) assessed on MRI | 5 years
  long-term secondary outcome
Changes in cerebral glymphatic function assessed by non-invasive diffusion tensor image analysis along the perivascular space (ALPS-index) | 6 months
  short-term secondary outcome
Changes in cerebral glymphatic function assessed by non-invasive diffusion tensor image analysis along the perivascular space (ALPS-index) | 2 years
  long-term secondary outcome
Changes in cerebral glymphatic function assessed by non-invasive diffusion tensor image analysis along the perivascular space (ALPS-index) | 5 years
  long-term secondary outcome
Changes in cerebral blood flow (CBF) in the territory of the culprit artery assessed by arterial spin labeling (ASL) perfusion image | 6 months
  short-term secondary outcome
Changes in cerebral blood flow (CBF) in the territory of the culprit artery assessed by arterial spin labeling (ASL) perfusion image | 2 years
  long-term secondary outcome
Changes in cerebral blood flow (CBF) in the territory of the culprit artery assessed by arterial spin labeling (ASL) perfusion image | 5 years
  long-term secondary outcome
Metabolite profiles in participants' faecal samples and serum samples | 6 months
  short-term secondary outcome: metabolite composition was analyzed via liquid chromatography tandem mass spectrometry (LC-MS/MS)
Metabolite profiles in participants' faecal samples and serum samples | 2 years
  long-term secondary outcome: metabolite composition was analyzed via liquid chromatography tandem mass spectrometry (LC-MS/MS)
Incidence of stroke event including ischemic and hemorrhagic stroke | 6 months
  short-term secondary outcome
Incidence of stroke event including ischemic and hemorrhagic stroke | 2 years
  long-term secondary outcome
Incidence of stroke event including ischemic and hemorrhagic stroke | 5 years
  long-term secondary outcome

IPD SHARING:
Plan to Share IPD: No